CLINICAL TRIAL: NCT04295252
Title: Cardiogenic Shock: a Prospective National Registry to Get Insights in Patients' Profile, Management and Outcome
Brief Title: Altshock-2 REGISTRY
Status: Recruiting | Type: Observational
Sponsor: Niguarda Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 45-12022020
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cardiogenic Shock
Keywords: cardiogenic shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cardiogenic shock patients: All-comers cardiogenic shock patients Admitted to the Intensive Coronary Care Units

SUMMARY:
The study will provide data on profile, management, outcome, and evolution over time of cardiogenic shock patients admitted to the Intensive Coronary Care Units

DETAILED DESCRIPTION:
Cardiogenic shock (CS) is the most severe form of acute heart failure. Data on epidemiology of CS have been drawn from previously published registries focussing on acute coronary syndrome (ACS) and myocardial infarction (AMI). Indeed, CS occurs in 5-7% of patients presenting with ACS and ACS has been reported as the most prevalent cause of CS, accounting for about 80% of cases.

However, recent evidences in a contemporary cohort in North America have shown that more than two-thirds of all cardiogenic shock cases were related to causes other than AMI and that these patients had outcomes at least as poor as patients with AMI-CS.

Given the high short-term mortality of these patients and the need for developing dedicated cardiac shock centres and systems of care to time our interventions, it is of utmost importance to achieve a better clinical phenotyping of the heterogeneous causes and presentations of CS patients and carefully perform research outcome.

Accordingly, the Altshock-2 registry will represent a unique opportunity to evaluate the full spectrum of CS admitted in Intensive Coronary Care Units and to collect a selected number of variables related to aetiology, clinical presentation, ongoing pharmacological treatments, use of mechanical support devices and outcome.

ELIGIBILITY:
All consecutive CS patients hospitalized in the above reported centres between January 2020 and December 2030.

Cardiogenic shock is defined as:

1. Systolic blood pressure (SBP) <90 mmHg or mean arterial pressure (MAP) <60 mmHg, after an appropriate fluid challenge if there is no sign of overt fluid overload, OR need of vasoactive agents to maintain SBP > 90 mmHg or MAP > 60 mmHg, OR need of MCS;
2. At least one of the following criteria/signs of overt hypoperfusion: mixed venous oxygen saturation <60%; arterial lactates > 2 mmol/L; oliguria < 0.5 ml/Kg/h for at least 6 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers cardiogenic shock patients admitted to the Intensive Coronary Care Units
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To provide data on profile, management, outcome, and evolution over time of CS patients admitted to ICCU | 10 years
  No formal sample size calculation was used to manage enrolment in the registry since the goal is to obtain participation by all possible eligible patients. No formal pre-specified hypothesis testing is planned. All analyses will be descriptive in nature Accordingly, measures of primary outcome will not be provided
Re-hospitalization | 10 years
  Number of patients

SECONDARY OUTCOMES:
To collect data on clinical characteristics and management of cardiogenic shock patients | 10 years
  Accordingly to the descriptive nature of the analyses, measures of secondary outcome will not be provided

CONTACTS AND LOCATIONS:
Locations (1):
- ASST GOM Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pagnesi M, Riccardi M, Sacco A, Viola G, Oliva F, Frea S, Briani M, Bertoldi LF, Bertaina M, Potena L, Valente S, Marini M, De Ferrari GM, D'Ettore N, Cardinale A, Camporotondo R, Rota M, Tavazzi G, Morici N, Pappalardo F, Metra M; Altshock-2 Investigators. Lactate Values and Mortality in Patients With Cardiogenic Shock: Insights From the Altshock-2 Registry. Crit Care Med. 2025 Aug 1;53(8):e1620-e1629. doi: 10.1097/CCM.0000000000006738. Epub 2025 Jun 12. PMID 40504883
- [Derived] Morici N, Frea S, Bertaina M, Sacco A, Corrada E, Dini CS, Briani M, Tedeschi M, Saia F, Colombo C, Rota M, Oliva F, Iannaccone M, De Ferrari GM, Sionis A, Kapur NK, Tavazzi G, Pappalardo F. SCAI stage reclassification at 24 h predicts outcome of cardiogenic shock: Insights from the Altshock-2 registry. Catheter Cardiovasc Interv. 2023 Jan;101(1):22-32. doi: 10.1002/ccd.30484. Epub 2022 Nov 15. PMID 36378673